CLINICAL TRIAL: NCT05756621
Title: SUPER-refractory Status Epilepticus After Cardiac Arrest: a Multicenter, Retrospective, Cohort Study of Dual Anti-glutamate Therapy With Ketamine and Perampanel
Brief Title: Dual Anti-glutamate Therapy in Super-refractory Status Epilepticus After Cardiac Arrest
Acronym: SUPER-CAT
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Collaborators: Azienda Ospedaliera San Gerardo di Monza (Other); Azienda Ospedaliero-Universitaria di Modena (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other); Ospedale Centrale Bolzano (Other); Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other); Azienda Ospedaliero-Universitaria Careggi (Other); Azienda Ospedaliero-Universitaria di Parma (Other); Santa Chiara Hospital (Other); Ospedale M. Bufalini Cesena (Other); Azienda Ospedaliera Brotzu (Other); Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Sponsor
Other Study IDs: SUPER-CAT
Record Dates: First submitted 2023-02-17; First posted 2023-03-06 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Status Epilepticus; Cardiac Arrest
Keywords: super-refractory; prognostic indicators; perampanel; ketamine
MeSH Terms: conditions — Status Epilepticus; Heart Arrest | interventions — Ketamine; perampanel; Levetiracetam; Valproic Acid; Phenytoin; Lacosamide; Topiramate; Propofol; Midazolam; Thiopental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Dual anti-glutamate therapy (DUAL): Patients who received ketamine as a continuous i.v. for 3 days (induction dose 1.5-3 mg/kg, followed by maintenance dose 2-10 mg/kg/h; dose adjustment according to EEG target of "ketamine pattern") + oral perampanel via nasogastric tube for 5 days (12 mg if weight > 60 kg; 9 mg if weight 50-60 kg; 6 mg if weight < 50 kg), followed by gradual dose reduction according to clinical evolution.
  Interventions: Drug: Ketamine
- Control (OTHERS): Patients who received any antiseizure and anesthetic therapy according to usual clinical practice, excluding the two anti-glutamate drugs ketamine and perampanel.
  Interventions: Drug: Any anti-epileptic and anesthetic therapy, excluding Ketamine and Perampanel

INTERVENTIONS:
Drug: Ketamine — "Dual anti-glutamatergic therapy" (DUAL) intervention group: patients who received ketamine as a continuous i.v. for 3 days (induction dose 1.5-3 mg/kg, followed by maintenance dose 2-10 mg/kg/h; dose adjustment according to EEG target of "ketamine pattern") + oral perampanel via nasogastric tube for 5 days (12 mg if weight > 60 kg; 9 mg if weight 50-60 kg; 6 mg if weight < 50 kg), followed by gradual reduction according to clinical evolution.
  Other Names: Perampanel
  Groups: Dual anti-glutamate therapy (DUAL)
Drug: Any anti-epileptic and anesthetic therapy, excluding Ketamine and Perampanel — Any antiseizure and anesthetic therapy according to usual clinical practice, excluding the two anti-glutamate drugs Ketamine and Perampanel
  Other Names: Levetiracetam, Valproate, Phenytoin, Lacosamide, Topiramate, Propofol, Midazolam, Thiopental
  Groups: Control (OTHERS)

SUMMARY:
Status epilepticus (SE) is found in 20-30% of patients in coma after cardiac arrest, is often refractory to medical therapy and is considered a negative prognostic factor. Intensity and duration of treatment of refractory and super-refractory post-anoxic SE pose the ethical dilemma between futility of treatments and, conversely, their premature suspension. A recent study by the Epilepsy Center of the San Gerardo Hospital has shown that patients with super-refractory post-anoxic SE and favorable prognostic indicators can achieve a good functional outcome in more than 40% of cases, if treated with intensive and protracted therapy.

However, there is profound uncertainty about the best combination of antiseizure medications and anesthetics to use in this condition. A combined anti-glutamatergic therapy with ketamine (anti-NMDA receptor) and perampanel (anti-AMPA receptor), aimed at counteracting the excitotoxicity linked to global cerebral ischemia, could be particularly effective in the treatment of super-refractory SE with post-anoxic etiology. Preliminary results in the first 26 patients treated in the Coordinating Center of the project indicate that this therapy appears safe and highly effective (80% SE resolution, 40% good neurological outcome).

The aim of the SUPER-CAT study is to investigate the efficacy and safety of combined therapy with ketamine and perampanel (dual anti-glutamatergic therapy) in patients with post-anoxic super-refractory status epilepticus, compared to other therapies, using a multi-centre, retrospective, cohort study design.

DETAILED DESCRIPTION:
Status epilepticus (SE) is found in 20-30% of patients in a coma after cardiac arrest, is frequently refractory to medical therapy and is usually considered a poor prognostic factor. The intensity and duration of treatment for post-anoxic refractory and super-refractory SE remains a highly controversial issue, posing the ethical dilemma between futility and premature discontinuation of care.

Although the TELSTAR randomized clinical trial demonstrated the futility of aggressive treatment in post-anoxic patients with generalized periodic pattern, the question remains open about the benefit of aggressive therapy in post-anoxic patients with SE properly defined according to the Salzburg criteria.

The latest guidelines of the European Resuscitation Council recommend the use of electroencephalogram (EEG) both for the neurological prognosis and for the diagnosis of post-cardiac arrest epileptic seizures, define the highly malignant EEG patterns (which do not include status epilepticus; while generalized periodic pattern and suppressed background are included) and recommend treatment of seizures with first-line antiepileptic therapy (levetiracetam or valproate), while there are no recommendations regarding second-line antiepileptic therapy. The same guidelines recommend a multi-modal approach, using different indicators (brainstem reflexes, somatosensory evoked potentials, EEG patterns, neuron-specific enolase [NSE] levels and neuroimaging) to arrive at the formulation of the neurological prognosis. A favorable neurological outcome is present in <15% of post-anoxic SE cases after moderate intensity treatment.

A recent study by the Epilepsy Center of the San Gerardo Hospital ASST Monza on a prospective cohort of 166 consecutive patients with cardiac arrest showed that patients with refractory post-anoxic SE and favorable prognostic indicators can achieve a good functional outcome (CPC 1-2) in > 40% of cases, if treated aggressively and prolonged with second-line anti-epileptic and anesthetic therapy.

However, there is profound uncertainty about the best combination of antiseizure medications and anesthetics to use in this condition. A pilot study of the Epilepsy Center of the San Gerardo ASST Monza hospital has shown an efficacy of 75% of anti-glutamatergic therapy with oral load of perampanel (anti-AMPA receptor), combined with different types of anesthetics (including ketamine, anti -NMDA receptor), in 8 patients with super-refractory post-anoxic SE. All patients included in this series presented the main favorable prognostic indicators (presence of brainstem reflexes, presence of N20 cortical evoked potentials, absence of generalized periodic pattern) and in 60% of cases (5 out of 8 cases) a neuroimaging with mild anoxic damage. The clinical outcome was favorable, with the achievement of functional independence in 50% of cases (4 cases out of 8) after 3 months.

A dual anti-glutamatergic therapy, performed by combining ketamine and perampanel could contrast in a particularly effective way the excitotoxicity linked to the global cerebral ischemia, favoring the resolution of the super-refractory SE and improving the global outcome of the post-cardiac arrest patient. Preliminary results in the first 26 post-anoxic super-refractory SE patients treated in the project Coordinating Center indicate that a dual anti-glutamatergic therapy with ketamine and perampanel appears highly effective (81% SE resolution; 41% good neurological outcome after 6 months) and without significant side effects. The selection of these patients was made on the basis of the multi-modal prognostic indicators described above, in accordance with the current guidelines on neurological prognosis.

The aim of the SUPER-CAT study is to evaluate the efficacy and safety of combined therapy with ketamine and perampanel (dual anti-glutamatergic therapy) in patients with super-refractory SE of post-anoxic aetiology, compared to other therapies, using a multi-centre, retrospective, cohort study design.

The study will be conducted thanks to the collaboration of the Intensive Care and Resuscitation Units and the Epilepsy Centers of 9 Italian hospitals, with the epidemiological-statistical coordination of the Mario Negri Institute for Pharmacological Research in Milan.

Patients with super-refractory status epilepticus after in-hospital or out-of-hospital cardio-circulatory arrest will be enrolled.

The results of the study will allow to compare the feasibility, efficacy and safety of dual anti-glutamate therapy with ketamine and perampanel in super-refractory post-anoxic SE compared to other anti-epileptic and anesthetic therapies used in normal clinical practice. If clinically relevant, these results will lay the foundations for the development of a subsequent randomized clinical trial.

The study has a retrospective observational design, therefore no interventions or modifications in conventional diagnostic and therapeutic procedures will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* patients in coma after cardio-circulatory arrest (CCA) admitted to the Intensive Care Unit and treated with target temperature management (TTM) for the first 24 hours
* initiation of continuous electroencephalographic (cEEG) monitoring within 24-36 hours of CCA
* diagnosis of super-refractory status epilepticus, relapsed after the first cycle of anesthetics (lasting > 24 hours) and antiepileptic therapy, defined according to the international Salzburg criteria9
* presence of pupillary reflex present bilaterally
* presence of N20 cortical response present bilaterally

Exclusion Criteria:

* EEG with periodic pattern (generalized periodic discharges; GPDs)
* status epilepticus resolved after the first cycle of anesthetics + antiepileptics
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with super-refractory status epilepticus after cardiac arrest, admitted to the Intensive Care Unit, with continuous EEG monitoring, presence of first-line favorable prognostic indicators (pupillary reflexes and N20 cortical responses bilaterally; absence of periodic EEG pattern).
  Outcomes will be also analyzed for the following pre-defined population:
  "Patients with favorable prognostic indicators": patients presenting 5 or more of the following: 1) presence of a pupillary reflex bilaterally; (2) presence of corneal reflex bilaterally; (3) presence of N20 cortical response bilaterally; (4) NSE <68 ng/mL at 24-72 hours from ACC; (5) absence of periodic EEG patterns (GPDs); (6) absence of severe anoxic brain damage on neuroimaging
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with resolution of status epilepticus | Over the entire period of stay in the Intensive Care Unit (up to 30 days)
  Number of patients with resolution of status epilepticus, not followed by relapse and without the use of additional antiepileptic drugs, evaluated over the entire period of stay in the Intensive Care Unit, in the two groups DUAL versus OTHERS

SECONDARY OUTCOMES:
Number of patients with with time-locked resolution of status epilepticus | first 5 days after start of therapy
  Number of patients with with resolution of status epilepticus 5 days after the start of therapy, not followed by relapse and without the use of additional antiepileptic drugs (only in the DUAL group)
Number of patients with early favorable neurological outcome | Over the entire period of stay in the Intensive Care Unit (up to 30 days)
  Number of patients with early favorable neurological outcome, defined as the patient's awakening (up to "command execution") during the stay in the Intensive Care Unit
Number of patients with favorable long-term neurological outcome | 6 months after cardiac arrest
  Number of patients with favorable long-term neurological outcome, defined by a modified Rankin scale score ≤ 2 at 6 months (minimum score 0, maximum score 6; lower scores indicate better outcomes)
mortality in intensive care | Over the entire period of stay in the Intensive Care Unit (up to 30 days)
  mortality in intensive care
mortality at 6 months | 6 months after cardiac arrest
  mortality at 6 months
cumulative probability of resolution of status epilepticus | Over the entire period of stay in the Intensive Care Unit (up to 30 days)
  incidence of the occurrence of resolution of status epilepticus, taking into account death as competing risk (cumulative incidence function)
Number of patients with abnormal cholestasis indices | Over the entire period of stay in the Intensive Care Unit (up to 30 days)
  Number of patients with abnormal cholestasis indices (GT-gamma > 3 times the upper limit of normal)
Number of patients with third degree atrioventricular block or cardiac arrest recurrence | Over the entire period of stay in the Intensive Care Unit (up to 30 days)
  Number of patients with third degree atrioventricular block or cardiac arrest recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Simone Beretta, MD, PhD, Principal Investigator — University of Milano Bicocca; Matteo Pozzi, MD, Study Chair — Fondazione IRCCS Gerardo dei Tintori Monza
Locations (10):
- Italy (10):
  - ASST Spedali Civili Brescia, Brescia, BS
  - Ospedale Centrale di Bolzano, Bolzano, BZ
  - Ospedale G. Brotzu, Cagliari, CA
  - Ospedale M. Bufalini, Cesena, FC
  - AOU Careggi, Florence, FI
  - Fondazione IRCCS San Gerardo dei Tintori Monza, Monza, MB
  - Azienda Ospedaliero-Universitaria di Modena, Modena, MO
  - Azienda Ospedaliero-Universitaria di Parma, Parma, PR
  - Ospedale Santa Chiara Trento, Trento, TN
  - Azienda Ospedaliero-Universitaria Integrata di Verona, Verona, VR

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mani R, Schmitt SE, Mazer M, Putt ME, Gaieski DF. The frequency and timing of epileptiform activity on continuous electroencephalogram in comatose post-cardiac arrest syndrome patients treated with therapeutic hypothermia. Resuscitation. 2012 Jul;83(7):840-7. doi: 10.1016/j.resuscitation.2012.02.015. Epub 2012 Feb 23. PMID 22366352
- [Background] Lybeck A, Friberg H, Aneman A, Hassager C, Horn J, Kjaergaard J, Kuiper M, Nielsen N, Ullen S, Wise MP, Westhall E, Cronberg T; TTM-trial Investigators. Prognostic significance of clinical seizures after cardiac arrest and target temperature management. Resuscitation. 2017 May;114:146-151. doi: 10.1016/j.resuscitation.2017.01.017. Epub 2017 Feb 3. PMID 28163232
- [Background] Cronberg T. Should Postanoxic Status Epilepticus Be Treated Agressively? Yes! J Clin Neurophysiol. 2015 Dec;32(6):449-51. doi: 10.1097/WNP.0000000000000209. PMID 26629753
- [Background] Dragancea I, Wise MP, Al-Subaie N, Cranshaw J, Friberg H, Glover G, Pellis T, Rylance R, Walden A, Nielsen N, Cronberg T; TTM trial investigators. Protocol-driven neurological prognostication and withdrawal of life-sustaining therapy after cardiac arrest and targeted temperature management. Resuscitation. 2017 Aug;117:50-57. doi: 10.1016/j.resuscitation.2017.05.014. Epub 2017 May 12. PMID 28506865
- [Background] Ruijter BJ, Keijzer HM, Tjepkema-Cloostermans MC, Blans MJ, Beishuizen A, Tromp SC, Scholten E, Horn J, van Rootselaar AF, Admiraal MM, van den Bergh WM, Elting JJ, Foudraine NA, Kornips FHM, van Kranen-Mastenbroek VHJM, Rouhl RPW, Thomeer EC, Moudrous W, Nijhuis FAP, Booij SJ, Hoedemaekers CWE, Doorduin J, Taccone FS, van der Palen J, van Putten MJAM, Hofmeijer J; TELSTAR Investigators. Treating Rhythmic and Periodic EEG Patterns in Comatose Survivors of Cardiac Arrest. N Engl J Med. 2022 Feb 24;386(8):724-734. doi: 10.1056/NEJMoa2115998. PMID 35196426
- [Background] Leitinger M, Trinka E, Gardella E, Rohracher A, Kalss G, Qerama E, Hofler J, Hess A, Zimmermann G, Kuchukhidze G, Dobesberger J, Langthaler PB, Beniczky S. Diagnostic accuracy of the Salzburg EEG criteria for non-convulsive status epilepticus: a retrospective study. Lancet Neurol. 2016 Sep;15(10):1054-62. doi: 10.1016/S1474-4422(16)30137-5. Epub 2016 Aug 8. PMID 27571157
- [Background] Nolan JP, Sandroni C, Bottiger BW, Cariou A, Cronberg T, Friberg H, Genbrugge C, Haywood K, Lilja G, Moulaert VRM, Nikolaou N, Mariero Olasveengen T, Skrifvars MB, Taccone F, Soar J. European Resuscitation Council and European Society of Intensive Care Medicine Guidelines 2021: Post-resuscitation care. Resuscitation. 2021 Apr;161:220-269. doi: 10.1016/j.resuscitation.2021.02.012. Epub 2021 Mar 24. PMID 33773827
- [Background] Dragancea I, Backman S, Westhall E, Rundgren M, Friberg H, Cronberg T. Outcome following postanoxic status epilepticus in patients with targeted temperature management after cardiac arrest. Epilepsy Behav. 2015 Aug;49:173-7. doi: 10.1016/j.yebeh.2015.04.043. Epub 2015 Jun 24. PMID 26117526
- [Background] Beretta S, Coppo A, Bianchi E, Zanchi C, Carone D, Stabile A, Padovano G, Sulmina E, Grassi A, Bogliun G, Foti G, Ferrarese C, Pesenti A, Beghi E, Avalli L. Neurologic outcome of postanoxic refractory status epilepticus after aggressive treatment. Neurology. 2018 Dec 4;91(23):e2153-e2162. doi: 10.1212/WNL.0000000000006615. Epub 2018 Oct 31. PMID 30381366
- [Background] Beretta S, Padovano G, Stabile A, Coppo A, Bogliun G, Avalli L, Ferrarese C. Efficacy and safety of perampanel oral loading in postanoxic super-refractory status epilepticus: A pilot study. Epilepsia. 2018 Oct;59 Suppl 2:243-248. doi: 10.1111/epi.14492. Epub 2018 Aug 29. PMID 30159874